CLINICAL TRIAL: NCT00474721
Title: A Randomized Blinded Comparison of Acetaminophen With Codeine and Ibuprofen for Treatment of Acute Pain in Children With Extremity Injuries
Brief Title: Comparison of Acetaminophen With Codeine and Ibuprofen for Children With Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCHSD10926
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Pain
Keywords: child; pain; analgesics
MeSH Terms: conditions — Pain | interventions — Ibuprofen; acetaminophen, codeine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ibuprofen
Drug: acetaminophen with codeine

SUMMARY:
We compared the pain relief of acetaminophen with codeine versus ibuprofen for children ages 5-18 years who came to the Pediatric Emergency Department with injuries to their arms or legs.

DETAILED DESCRIPTION:
We conducted a randomized, double-blinded equivalence trial. Pediatric Emergency Department patients 5-18 years of age with acute extremity pain received acetaminophen-codeine (1 mg/kg as codeine) or ibuprofen (10 mg/kg). They provided Color Analog Scale pain scores at baseline and at 20, 40, and 60 minutes after medication administration. The primary outcome measured was the difference in changes in pain score at 40 minutes, compared against a previously described minimal clinically significant change in pain score of 2 cm. Additional outcomes included need for rescue medication and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 18 years of age
* Spoke English as a primary language
* Complained of an extremity injury with tenderness to palpation from the clavicle or femoral neck to the distal phalanges
* Scored 5 or greater on a 10-point ordinal or Varni-Ryan pain scale administered at triage

Exclusion Criteria:

* Allergy or prior adverse reaction to acetaminophen, codeine or ibuprofen;
* Administration of any analgesic within 6 hours of presentation;
* Significant deformity or vascular insufficiency of the extremity requiring immediate treatment as determined by the treating physician;
* Inability to use the study pain instrument;
* Any laceration near the suspected injury;
* Chronic hepatic or renal disease;
* Pregnancy in the third trimester;
* Concurrent use of contraindicated medications such as monoamine oxidase inhibitors; or
* Use of central nervous system depressants such as ethanol, benzodiazepines, barbiturates, antidepressants, or recreational drugs

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2002-11; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Change in color analog scale pain score | 40 minutes

SECONDARY OUTCOMES:
adverse reaction | during ED stay
need for rescue medication | during ED stay
Change in pain score | 20 and 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Janet H Friday, Principal Investigator — UCSD, Dept of Pediatrics and Rady Children's Hospital
Locations (1):
- Rady Children's Hospital, San Diego, California, United States